CLINICAL TRIAL: NCT01820728
Title: A Phase III Clinical Study for the Comparison Evaluation of DA-3801 and Gonal-F® in Infertile Female Patients With Chronic Anovulation Syndrome
Brief Title: A Phase III Clinical Study to Compare the Efficacy and Safety of DA-3801 and That of Gonal-F®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA3801_CA_III (Version 5.1)
Record Dates: First submitted 2013-03-18; First posted 2013-03-29 (Estimated); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Infertility; Anovulation
MeSH Terms: conditions — Infertility; Anovulation | interventions — DA-3801; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DA-3801 injection (Experimental): Recominant human follicle stimulating hormone 75 IU/day is injected for 14 days
  Interventions: Drug: DA-3801 Injection
- Gonal-F® (Active Comparator): 75 IU/day is injected for 14 days
  Interventions: Drug: Gonal-F®

INTERVENTIONS:
Drug: DA-3801 Injection
  Arms: DA-3801 injection
Drug: Gonal-F®
  Arms: Gonal-F®

SUMMARY:
open label, active-controlled, randomized, parallel group, comparative study.

DETAILED DESCRIPTION:
This is a phase III comparative study to evaluate the effectiveness and safety of DA-3801 in treatment of the patients with WHO Group II anovulatory infertility failing to clomiphene citrate treatment. The study is conducted with following methods: open label, active-controlled, randomized, parallel group, comparative.

ELIGIBILITY:
Inclusion Criteria:

* WHO group II
* Clomiphene citrate resistance
* BMI: 17~29 kg/m^2
* Irregular menstrual cycle
* Normal blood concentration of FSH, E2, prolactin and TSH

Exclusion Criteria:

* Uncontrolled endocrine disease
* Ovarian cystic tumor which are NOT related to PCOS
* Severe endometriosis
* Chronic cardiovascular disease, liver complaint

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2007-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The ovulation rate after 3 cycles of the injection | 5 weeks maximum

SECONDARY OUTCOMES:
Total dose used, IU (International Unit) | 5 weeks
Duration of stimulation, days | 5 weeks
Threshold dose, IU | 5 weeks
Number of follicles | 5 weeks
  Counter the number of follicles which are 12 mm, 15 mm, 18 mm in diameter

CONTACTS AND LOCATIONS:
Overall Officials: Eung Gi Min, M.D., Ph.D., Principal Investigator — Dongguk University Hospital; Chang Suk Suh, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital; Doo Seok Choi, M.D., Ph.D., Principal Investigator — Samsung Medical Center; Chung Hoon Kim, M.D., Ph.D., Principal Investigator — Asan Medical Center; Jong Min Park, M.D.,Ph.D., Principal Investigator — Gachon University Gil Medical Center; Kyung Joo Hwang, M.D., Ph.D., Principal Investigator — Ajou University School of Medicine
Locations (1):
- Seoul National University Hospital Institutional Review Board, Seoul, South Korea